CLINICAL TRIAL: NCT00599001
Title: A Phase 1, Randomized, Single-Blind, Placebo-Controlled Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of SD-101 in Healthy Normal Male Volunteers
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of SD-101 in Healthy Normal Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DV3-HNV-01
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: healthy volunteer; research subjects; Immunostimulatory sequence (ISS); phase 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escalating Dose of SD-101 (Experimental)
  Interventions: Drug: SD-101
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SD-101 — Single subcutaneous escalating dose
  Arms: Escalating Dose of SD-101
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the safety, tolerability, and biological activity of SD-101 compared with placebo in healthy male volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, single-blind, placebo-controlled study of five escalating dose levels of SD-101 in healthy male volunteers. The objectives of the study are to assess the safety, tolerability, pharmacokinetic profile, and pharmacodynamics of SD-101. Approximately 40 subjects will participate.

Once subjects have been consented, screened, and assigned to one of the dose levels of SD-101, subjects will receive a single subcutaneous injection of either SD-101 or placebo (PBS) in a ratio of 6:2.

Safety and tolerability will be evaluated by occurrence of adverse events, blood and urine laboratory tests, physical examination findings, vital signs , and electrocardiogram findings. Pharmacodynamics will be evaluated by levels of blood biomarkers and serum cytokines, and flow cytometric cell counts. Pharmacokinetics will be evaluated by levels of study drug in serum.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written, informed consent must be obtained from the subjects before any study-specific procedures are performed.
* Subject must be male and 18 years of age or older.
* Subject must be willing to submit to a urine drug screen and agree to abstain from alcohol, caffeine, and tobacco during the required stay in the Phase I Unit.
* Subject must be willing to abide by the rules of the Phase 1 Unit.
* Subjects whose sexual partners are of childbearing potential must agree to use an effective method of birth control (i.e., chemical contraceptives, barrier plus spermicide, intrauterine device) during the treatment phase and for 14 days post treatment.
* Must be negative for Hepatitis B and C and human immunodeficiency virus (HIV).

Exclusion Criteria:

* Females.
* Clinically significant active, acute, or chronic illness.
* History of coagulation or bleeding disorders.
* Clinically significant chronic or recent (within 21 days of dosing) acute gastrointestinal disorder with nausea, vomiting or diarrhea as a major symptom.
* Received any vaccine within 3 weeks of study entry or plans to be vaccinated within 6 weeks after study injection.
* History of significant cardiovascular or cerebrovascular disease.
* History of evaluation for autoimmune disease including systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), scleroderma or thyroiditis.
* Significant psychiatric illness that could potentially interfere with the assessments during this study.
* Subjects who have had prior surgery or a major infection within 6 months of dosing.
* History of medications within 7 days of dosing, except vitamins and/or minerals.
* History of Gilbert's disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with and the amplitude and timing of adverse events, proportion of subjects with and the grade and timing of abnormal lab values, and proportion of subjects with and timing of changes in physical exam findings and vital signs | Up to 7 days after dosing

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Up to 24 hours after dosing
Levels of serum cytokines | Up to 7 days after dosing
Levels of blood biomarkers (interferon-alpha inducible genes) | Up to 7 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ruff, MD, Principal Investigator — Healthcare Discoveries, Inc.
Locations (1):
- Healthcare Discoveries, Inc., San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
No Change to status of this study.

REFERENCES:
- See also: Sponsor Website — http://www.dynavax.com